CLINICAL TRIAL: NCT07368049
Title: MR 7700 Multinuclear Application Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 301455
Record Dates: First submitted 2025-11-24; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma; MRI
Keywords: HCC; multinuclear; MR; Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCC patients (Experimental): HCC patients
  Interventions: Device: MR Scanning with Phosphorus nucleus + Sodium nucleus
- Healthy volunteers (Placebo Comparator): Healthy volunteers
  Interventions: Device: MR Scanning with Phosphorus nucleus + Sodium nucleus

INTERVENTIONS:
Device: MR Scanning with Phosphorus nucleus + Sodium nucleus — Using the Magnetic Resonance Equipment to perform phosphorus nucleus (31P) and sodium nucleus (23Na) scanning

SUMMARY:
The purpose of this clinical study is to perform phosphorus nucleus (31P) and sodium nucleus (23Na) imaging of the liver in patients with primary hepatocellular carcinoma (HCC) and healthy volunteers using the MR 7700 Magnetic Resonance Equipment, in order to explore the manifestations of multinuclear imaging in HCC patients and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 1. HCC patient group

  * Age ≥ 18 years;
  * With clear consciousness, ability to cooperate, and autonomous behavior;
  * Voluntary agreement to participate in this clinical trial and signing of the subject's informed consent form;
  * Patients diagnosed with primary hepatocellular carcinoma by imaging or clinical diagnosis, and who have not received tumor treatment.
* 2. Healthy control group

  * Age ≥ 18 years;
  * With clear consciousness, ability to cooperate, and autonomous behavior;
  * Voluntary agreement to participate in this clinical trial and signing of the subject's informed consent form;
  * No previous history of liver disease.

Exclusion Criteria:

* HCC patient group and healthy control group

  * Patients with claustrophobia.
  * Subject's body temperature > 39.5°C on the day of scanning.
  * Females who plan to be pregnant within 6 months, and pregnant and lactating females.
  * Patients with other implants, prostheses, foreign bodies, patches, etc. that are not suitable for MRI examination; patients with electronic implants, such as pacemakers, stimulators, insulin pumps, cochlear implants, etc.
  * Critically ill subjects with various resuscitation devices or those with any emergency medical condition requiring first aid.
  * Subjects with poor compliance are considered to be excluded by the investigators.
  * Subjects who are not considered suitable for this trial by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Ratio of metabolites （PME/PDE） | 14 days (anticipated)] after finishing 31P-MRS scanning
  By comparing the ratios of metabolites (PME/PDE) in the liver, the effectiveness of 31P magnetic resonance spectroscopy (31P-MRS) was evaluated.
  Theoretically,the PME/PDE ratio in patients with HCC was higher than that in healthy volunteers.
Image quality of 23Na-MRI | 14 days (anticipated)] after finishing 23Na-MRI scanning
  Image quality will be assessed by Likert score (1-5)
Adverse Event | From the time the subjects signed the ICF to completion of study visit(1 day).
  Monitor adverse events and serious adverse events during the study,summarize and analyze the frequency and percentage of all adverse events (including severe adverse events)

IPD SHARING:
Plan to Share IPD: Undecided